CLINICAL TRIAL: NCT04224142
Title: An Observational Study to Evaluate Metabolic Control and Dietary Management in Women With PKU Taking PKU Sphere During Pre-conception and/or Pregnancy
Brief Title: Evaluation of PKU Sphere in Maternal PKU
Acronym: Maternal PKU
Status: Completed | Type: Observational
Sponsor: Vitaflo International, Ltd (Industry)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: MCT-GMP-2018-08-14; 256857 (Other: IRAS); 19/NW/0167 (Other: HRA)
Record Dates: First submitted 2019-10-07; First posted 2020-01-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Maternal Phenylketonuria
Keywords: Maternal; PKU; Phenylketonuria; GMP; Glycomacropeptide
MeSH Terms: conditions — Phenylketonuria, Maternal; Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PKU sphere: PKU sphere (an FSMP) as per individual requirements determined by a dietitian.
  Interventions: Dietary Supplement: PKU sphere

INTERVENTIONS:
Dietary Supplement: PKU sphere — PKU sphere is a Food for Special Medical Purposes (FSMP). This product is for use in the dietary management of phenylketonuria (PKU).
  It is a powdered, low phenylalanine medical food containing a balanced mix of GMP, essential and non-essential amino acids, carbohydrate, fat, vitamins, minerals, and DHA.
  It is available in 27g sachets providing 15g PE and contains 28mg Phe and 35g sachets providing 20g PE and contains 36mg Phe.

SUMMARY:
This observational study aims to recruit females, aged 16 years and over, with phenylketonuria (PKU) or hyperphenylalaninemia (hyperphe) following dietary management advice pre-conception and/or during pregnancy, who are willing to take PKU sphere as part of their dietarty management.

DETAILED DESCRIPTION:
The aim of this study is to observe dietary management and metabolic control in women taking PKU sphere pre-conceptually and/or during pregnancy. To do this the following data points will be captured:

* Blood spot phenylalanine and tyrosine levels to measure metabolic control
* Changes to dietary management and any adaptations arising from incorporating PKU Sphere
* Compliance/adherence of patients to their recommended amount of protein substitute prescription.
* Tolerance of PKU sphere with respect to gastrointestinal (GI) symptoms and pregnancy associated nausea and vomiting.
* Acceptability of concurrent protein substitute(s) (if applicable).
* Nutritional status and weight management.
* Routine standard of care data on the final pregnancy outcome and postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of phenylketonuria (PKU) or hyperphenylalaninemia (hyperphe) which requires dietary management during pre-conception and/or pregnancy.
* Aged 16 years and above.
* Following dietary management advice pre-conceptually and/or during pregnancy, aiming for phenylalanine levels of 120-250µmol/L.
* Prior positive PKU sphere taste test completed as part of routine care.
* Chosen to take part or full requirement of protein substitute as PKU sphere pre-conceptually and/or during pregnancy.
* Willingly given, written, informed consent from patient.
* Participant is, in the opinion of the investigator, able to participate and can comply with the study protocol.

Exclusion Criteria:

* Conception of pregnancy without commencement of phe-restricted diet and blood phenylalanine not maintained within target range by 10 weeks' gestation.
* Patients with known soya, milk or fish allergies / intolerance.
* Intake of pegvaliase or large neutral amino acids within 30 days prior to screening visit.
* Patients who are currently participating in, plan to participate in, or have participated in an interventional investigational drug, food or medical device trial within 30 days prior to screening visit.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Maternal and preconception females, aged 16 years onwards with phenylketonuria (PKU) requiring dietary management with protein substitutes.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Change in blood spot phenylalanine levels | Baseline, 1-2 times weekly during preconception (max. 2 years), 2-3 times weekly during pregnancy, one month postpartum.
  Measurement of fasting phenylalanine concentrations completed once (1) to twice (2) weekly preconception (which may last for an indeterminate amount of time), twice (2) to three (3) times weekly during pregnancy and one month postpartum. Collected as dried bloodspots on Guthrie cards in the patient's own home and posted to the hospital laboratory for analysis.
Change in blood spot tyrosine levels | Baseline, 1-2 times weekly during preconception (max. 2 years), 2-3 times weekly during pregnancy, one month postpartum.
  Measurement of fasting tyrosine concentrations completed once (1) to twice (2) weekly preconception (which may last for an indeterminate amount of time), twice (2) to three (3) times weekly during pregnancy and one month postpartum. Collected as dried bloodspots on Guthrie cards in the patient's own home and posted to the hospital laboratory for analysis.
Change in adherence to study product intake | Every 12 weeks from baseline during preconception (max. 2 years) and pregnancy until the end of the pregnancy
  3-day diary recording compliance/adherence of patients to their prescribed amount of protein substitute.
Participants' gastrointestinal adverse events | Throughout the study until one month postpartum
  Participant to report any gastrointestinal (GI) symptoms and pregnancy-associated nausea and vomiting while consuming PKU Sphere.
Change in weight | Baseline, every 24 weeks during preconception (max. 2 years) and pregnancy, one month postpartum
  Weight (kg)
Change in plasma amino acid profile | Baseline, all routine results during preconception (max. 2 years) and pregnancy, one month postpartum
  Plasma amino acid profile
Change in plasma micronutrient profile | Baseline, all routine results during preconception (max. 2 years) and pregnancy, one month postpartum
  Plasma micronutrient profile
Pregnancy outcome | End of pregnancy
  Standard of care data on the outcome of the pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Ellerton, Principal Investigator — University College London Hospitals
Locations (3):
- United Kingdom (3):
  - Royal Victoria Hospital, Belfast
  - University Hospital of Wales, Cardiff
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No